CLINICAL TRIAL: NCT02200874
Title: Investigation of the Effectiveness and Efficiency of a Structural Clinical Nutrition Support by an Interdisciplinary Nutrition Support Team at the University Hospital Tübingen
Brief Title: Investigation of the Effectiveness and Efficiency of a Structural Clinical Nutrition Support
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Hohenheim (Other)
Collaborators: Center for Nutritional Medicine Tuebingen/Hohenheim (Unknown); University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Stephan C. Bischoff, MD, Professor, Prof. Dr., University of Hohenheim
Other Study IDs: ZEM_NST_KET
Record Dates: First submitted 2014-07-23; First posted 2014-07-25 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Malnutrition
Keywords: disease related malnutrition; influence of Nutrition Support Team; length of hospital stay; quality of life; body composition; health care costs
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- before NST-implementation (group A): Patients with a NRS of 3 or more than 3 or NUTRIC score of 4 or more than 4 within the first three days after admittance to hospital. Time point: Before implementation of Nutrition Support Team (NST).
- After NST-implementation (group B): Patients with a NRS of 3 or more than 3 or NUTRIC score of 4 or more than 4 within the first three days after admittance to hospital. Time point: After implementation of Nutrition Support Team (NST).

SUMMARY:
The purpose of this study is to investigate the effectiveness and efficiency of a structural clinical nutrition support by an interdisciplinary Nutrition Support Team. To do this we examine nutritional management and its economic impact as well as the nutritional status of patients of University Hospital Tübingen before and after the implementation of a Nutritional Support Team.

DETAILED DESCRIPTION:
In German hospitals disease related malnutrition is a major problem. Malnutrition is known to be associated with decreased quality of life, altered body composition as well as increased length of hospital stay. Guidelines recommend the installation of Nutrition Support Teams (NST) to combat this situation. However, the majority of German hospitals lacks a NST.

In the present study, we want to examine the effectiveness and efficiency of a Nutrition Support Team (NST) in an University hospital with 1500 beds. To do this we investigate the nutritional management, its economic impact and patient related data before and after NST-implementation. Examinations include a structural analysis of the hospital with regard to nutritional procedures and a patient-based analysis.

Patients are recruited from three representative normal wards and two intensive care units. Here we identify patients with risk for malnutrition with the help of nutritional screening tools (NRS 2002 [Nutritional Risk Screening]; NUTRIC [Nutritional Risk in the critically ill] Score).This is performed within the first three days after admittance. The patients with risk for malnutrition (NRS 2002 of 3 or more than 3, NUTRIC Score of 4 or more than 4) are included for further investigations. These include anthropometric measurements , assessment of body composition, evaluation of nosocomial infection and decubitus rate, quality of life (SF-12 questionnaire), length of hospital stay, evaluation of mortality risk, organ function and severity of illness as well as economic factors. Most examinations are repeated weekly depending from the length of stay in hospital.

All this examinations and evaluations will be collected at two time points. Before and after the implementation of a nutritional support team. That means we have two groups: group A- before NST-implementation (n=420) and group B - after NST-implementation (n=420).

After the whole data collection we want to compare the results of the two groups.

ELIGIBILITY:
Inclusion Criteria:

* patient of University Hospital Tübingen
* patient of one of the study-wards: Gastroenterology, Otolaryngology, Visceral and transplantation surgery, Internal intensive care unit, Surgery intensive care unit
* written informed consent of the patient/advisor
* risk of malnutrition: NRS Score of 3 or more than 3, NUTRIC Score of 4 or more than 4

Exclusion Criteria:

* age under 18 years
* withdrawn of written informed consent
* length of hospital stay shorter than 2 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from University Hospital Tübingen. 420 patiens in each group. Patients from three general wards and two intensive care units. From all patients written informed consent is needed. From sedated and/or ventilated patients, consent from their advisor is needed.
Sampling Method: Non-Probability Sample
Enrollment: 840 (Estimated)
Dates: Start 2012-11; Primary Completion 2016-12 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
length of hospital stay | Patients will be followed for the duration of hospital stay. Average hospital stay is about 7 days.

SECONDARY OUTCOMES:
case-related total costs of length of hospital stay | At time of hospital discharge.Average hospital stay is about 7 days.
Score (points) of Nutritional risk Screening | Within the first 3 days after admittance
  Patients at normal wards are screened with NRS 2002 (Nutritional Risk Screening 2002). Patients at intensive care units are screened with NUTRIC (Nutritional Risk in the critically ill) Score.
Score (points) of Nutritional risk Screening | Every 7th day after admittance- until discharge. Average hospital stay is about 7 days.
  Patients on normal wards are screened with NRS 2002 (Nutritional Risk Screening 2002). Patients on intensive care units are screened with NUTRIC (Nutritional Risk in the critically ill) Score.
  The screening is repeated weekly.

OTHER OUTCOMES:
body composition | Within the first 3 days after admittance
  To measure the body composition we use the bioelectrical impedance analysis. We evaluate the phase angle and ECM (extracellular cell mass)/BCM (body cell mass) ratio.
case-individual costs of hospital stay | At time of hospital discharge.Average hospital stay is about 7 days.
BMI | Within the first 3 days after admittance
  To asses the BMI we measure the height and weight of the patients and calculate the BMI.
body composition | Every 7th day after admittance -until discharge. Average hospital stay is about 7 days.
  To measure the body composition we use the bioelectrical impedance analysis. We evaluate the phase angle and ECM (extracellular cell mass)/BCM (body cell mass) ratio.
mortality risk | Within the first 3 days after admittance
  We evaluate the mortality risk by using SAP II (Simplified Acute Physiology) Score. The SAP II Score is only used on patients at intensive care units.
severity of illness and organ function | Every day -from first day of hospital stay to discharge.Average hospital stay is about 7 days.
  We evaluate the severity of illness and organ function by using SOFA (Sequential Organ Failure Assessment) Score. The SOFA Score is only used on patients at intensive care units.
decubitus risk | within the first 3 days after admittance
  We evaluate decubitus-risk by using Braden-Scale.
decubitus risk | Every 7th day after admittance- until discharge. Average hospital stay is about 7 days.
  We evaluate decubitus-risk by using Braden-Scale.
nosocomial infection | At time of hospital discharge.Average hospital stay is about 7 days.
quality of life | within 3 days after admittance
  Quality of life is assessed by using the standardized questionnaire "short-form" 12 ( SF-12).
quality of life | Every 7th day after admittance -until discharge. Average hospital stay is about 7 days.
  Quality of life is assessed by using the standardized questionnaire "short-form 12" (SF-12).
mortality | From day 1 to discharge.Average hospital stay is about 7 days.
BMI | Every 7th day after admittance -until discharge. Average hospital stay is about 7 days.
  To asses the BMI we measure the height and weight of the patients and calculate the BMI.
  The calculation is repeated weekly.

CONTACTS AND LOCATIONS:
Overall Officials: Stephan C. Bischoff, Professor, Study Director — Departement of Nutritional Medicine, University of Hohenheim, Stuttgart, Germany
Locations (1):
- University Hospital of Tübingen, Tübingen, Germany

REFERENCES:
- [Derived] Gonzalez-Granda A, Schollenberger A, Thorsteinsson R, Haap M, Bischoff SC. Impact of an interdisciplinary nutrition support team (NST) on the clinical outcome of critically ill patients. A pre/post NST intervention study. Clin Nutr ESPEN. 2021 Oct;45:486-491. doi: 10.1016/j.clnesp.2021.06.018. Epub 2021 Jun 26. PMID 34620359